CLINICAL TRIAL: NCT04223882
Title: Stress Management in Patients With Coronary Artery Disease: a Randomized Clinical Trial
Brief Title: Stress Management in Patients With Coronary Artery Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UP 5648/19
Record Dates: First submitted 2020-01-08; First posted 2020-01-10 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Stress, Psychological
Keywords: Stress, Psychological;; Coronary Artery Disease;; Percutaneous Coronary Intervention;; Endothelium;
MeSH Terms: conditions — Stress, Psychological; Coronary Artery Disease

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Intervention- Management of stress (Experimental): Patients in the intervention group will receive usual medical care and more stress management intervention. Stress management with cognitive behavioral techniques will be implemented one month after hospital discharge in the intervention group. Group sessions will be held between 6-9 people. There will be 3 1-hour meetings for 3 weeks. The intervention will be performed by psychologist.
  Interventions: Behavioral: Management of Stress
- Group Control (Active Comparator): Patients in the control group will receive usual medical care.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Management of Stress — Psychoeducation:
  Coronary artery disease, Percutaneous Coronary Intervention, traditional risk factors and emotional stress.
  Stress: physiology, triggers, triad (thinking, emotion, action).
  Skills training:
  Identify warning signs - signs and symptoms; Monitoring of irrational automatic thoughts generating alternative interpretations of situations or unrealistic thinking patterns (Dysfunctional Thinking Records Sheet).
  Self-control for stress management:
  Assertiveness training, problem solving. Thought-stopping technique, designed for dysfunctional thoughts, such as, "I won't do it," "It won't work."
  Stress Relief / Control Techniques:
  Diaphragmatic Breathing: Expansion of the abdomen rather than the chest when breathing.
  Progressive Muscle Relaxation: Maximize tension and alternately relax the muscles (legs, abdomen, chest, arms and face).
  Arms: Group Intervention- Management of stress
Other: Usual care — outpatient medical appointments
  Other Names: Patients in the control group will receive usual medical care
  Arms: Group Control

SUMMARY:
Introduction: Stress can cause hemodynamic and metabolic changes that contribute to endothelial dysfunction and there is a significant association between high stress and cardiovascular events. Objective: To evaluate the influence of stress management on endothelial function in patients undergoing percutaneous coronary intervention (PCI). Methods: Randomized, controlled, parallel, intention-to-treat clinical trial. Will be considered eligible patients who underwent percutaneous coronary intervention and who have high stress (above average for the Brazilian population) in the Perceived Stress Scale (PSS-10). Patients will be evaluated on PCI admission and stress management with cognitive behavioral techniques will be implemented one month after hospital discharge in the intervention group. Group sessions will be held between 6-9 people. There will be 4 1-hour meetings for 8 weeks. The primary outcome will be the difference in the variation of brachial artery flow-mediated dilatation (FMD) between the groups and at 3 months of baseline evaluation and at 6-month follow-up after the intervention and the secondary outcome will be the difference in the variation of the velocity of brachial artery. Pulse wave evaluated at the same time periods as DMF. Outcomes will be evaluated by Generalized Estimation Equations (GEE). Expected Results: In patients undergoing high-stress percutaneous coronary intervention, the use of cognitive behavioral techniques for stress management will improve endothelial function and vascular stiffness.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* Patients with CAD - obstruction of one or more epicardial arteries with at least 70% stenosis and / or Left Coronary Trunk (TBI) with at least 50% - measured by catheterization (CATE) and having performed elective PCI
* High stress: above average score for the Brazilian population in the Perceived Stress Scale (PSS-10)
* Signing of the Informed Consent.

Exclusion Criteria:

* Age ≥ 80 years
* Patients with inpatient events (AMI, CABG, stroke)
* Indication of catheterization for valvulopathies or congenital heart disease
* Severe aortic stenosis / Ejection fraction <30%, cardiomyopathy, severe congestive heart disease
* Severe diseases with life expectancy <6 months
* Cognitive or mental difficulties to understand the instrument
* Inability to follow up visits

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-10-05 (Actual); Primary Completion 2023-01-05 (Actual); Study Completion 2023-10-05 (Estimated)

PRIMARY OUTCOMES:
Difference in Flow-mediated Dilation in the Brachial Artery in the Base and After the Treatment. | Three months after the first evaluation
  Inter group difference in flow-mediated dilation in the brachial artery in the baseline and after the treatment (about Three months after the first).
  Vasodilatation of the endothelium-dependent brachial artery was evaluated by ultrasound using a 3-12 MHz linear transducer. Three images of the basal diameter (BD) of the brachial artery at the end of the diastole were acquired, as well as the mean velocity of the baseline arterial flow, with the linear transducer positioned 5 cm above the antecubital fossa. Subsequently, the sphygmomanometer was placed in the arm and inflated 50 mmHg above baseline systolic blood pressure for five minutes. After that, 3 images of the arterial diameter were acquired up to 80 seconds of the deflation of the cuff (post-occlusion diameter- PD), as well as the average of the arterial flow velocity. Flow-dependent vasodilation responses were expressed as a percentage variation from the baseline brachial diameter (PD-BD/ BD x 100).

CONTACTS AND LOCATIONS:
Overall Officials: Marcia Moura Schmidt, PhD, Study Director — Instituto de Cardiologia do Rio Grande do Sul; Karine Elisa Schwarzer Schmidt, Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Marcia Moura Schmidt, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No